CLINICAL TRIAL: NCT05923138
Title: aBOrdaje nutriCional en ADultos Seguidos en hOspitales eSpañoles Por Insuficiencia Cardiaca (BOCADOS-IC)
Brief Title: Nutritional Approach in Adults Followed up in Spanish Hospitals for Heart Failure (BOCADOS-IC)
Acronym: BOCADOS-IC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, JOSE ANGEL PEREZ RIVERA, Principal Investigator, Spanish Society of Cardiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEC-BOCADOS-IC-2023; SECAINC-INV-ICC 23/04 (Other: SOCIEDAD ESPAÑOLA DE CARDIOLOGIA)
Record Dates: First submitted 2023-06-09; First posted 2023-06-28 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
Keywords: HEART FAILURE; MALNUTRITION
MeSH Terms: conditions — Heart Failure; Malnutrition | interventions — Exercise; Dietary Supplements

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NUTRITIONAL INTERVENTION (Experimental)
  Interventions: Dietary Supplement: MULTIDOMAIN NUTRITIONAL INTERVENTION: DIET, EXERCISE AND NUTRITIONAL SUPPLEMENTS
- CONTROL (Placebo Comparator)
  Interventions: Dietary Supplement: CONTROL

INTERVENTIONS:
Dietary Supplement: MULTIDOMAIN NUTRITIONAL INTERVENTION: DIET, EXERCISE AND NUTRITIONAL SUPPLEMENTS — Nutritional intervention (diet, dietetic recommendations and/or supplements). Participants will receive specific recommendations about diet, energetic dietetic supplementation, oral nutritional supplements, exercise... The "Nutrition Team" (formed by cardiologists, dieticians, nurses...) will closely monitor patients with periodic visits and reassessment of nutritional status and compliance with recommendations.
  Other Names: NUTRITION TEAM
  Arms: NUTRITIONAL INTERVENTION
Dietary Supplement: CONTROL — Standard treatment (usual recommendations in patients with heart failure)
  Arms: CONTROL

SUMMARY:
This is a randomized, controlled, open-label, prospective, multicentre clinical trial designed to assess the effects of a nutritional intervention on morbidity and mortality in patients with chronic heart failure.

Through a simple 1:1 randomization process, patients will be assigned to the control group or the intervention group. Patients in the intervention group will undergo an individualised nutritional intervention program consisting of 3 pillars: diet optimization, specific recommendations ,and nutritional supplementation if nutritional targets are not achieved.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 65 years with malnutrition (MNA-SF score ≤ 11) with chronic ambulatory heart failure (HF).

Exclusion Criteria:

* Admission for heart failure (HF) in the last month,
* Chronic renal failure on dialysis.
* Patients already on nutritional treatment.
* Concomitant diseases which, apart from the HF itself, could lead to a life expectancy of less than 1 year,
* Patients included in other clinical trials.
* Patients whose clinical situation makes it impossible to perform a nutritional assessment according to the design established in the study protocol or who do not give their consent for this purpose.
* Patients who during admission undergo surgical or percutaneous treatment to correct the cause of acute HF,

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
COMBINED EVENT | 6 MONTHS
  Time to the combined event of all-cause mortality or admission for heart failure at 6 months

SECONDARY OUTCOMES:
Time to 6-month cardiovascular mortality | 6 MONTHS
Time to all-cause admission at 6 months | 6 MONTHS
Changes in quality of life at 3 and 6 months post-intervention | 6 MONTHS
  Changes in the scores of Minnesota living with heart failure questionnaire
Changes in nutritional status at 3 and 6 months post intervention | 6 MONTHS
  Changes in the scores of Mini Nutritional Assessment Short Form

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No